CLINICAL TRIAL: NCT01203995
Title: Remote Information Counseling for Elders
Acronym: RICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kimberly Hemmerlein, Research Coordinator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0710-65B
Record Dates: First submitted 2010-09-01; First posted 2010-09-17 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Nutrition Assessment; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Usual Care (No Intervention)
- brief nutrition education (Experimental)
  Interventions: Behavioral: Nutrition information
- In Center training (Active Comparator)
  Interventions: Behavioral: Nutrition education and exercise training
- Video Conference training (Experimental)
  Interventions: Behavioral: Nutrition education and exercise training

INTERVENTIONS:
Behavioral: Nutrition information — Brief nutrition education with take home reference materials and portion size tools
  Arms: brief nutrition education
Behavioral: Nutrition education and exercise training — Twice per week nutrition education and exercise class held either in-clinic or through vide-conference.
  Arms: In Center training; Video Conference training

SUMMARY:
The purpose of this study is to provide testing methods of delivering nutrition and physical activity services for weight loss.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40 to 64 years.
2. One or more CHC visits in the past 12 months.
3. Body-mass index of ≥30 and <50.
4. English speaking.
5. Access to telephone.
6. A permanent address.
7. Willingness to be randomized.
8. Willingness to have computer installed in home.

Exclusion Criteria:

1. Any serious medical condition likely to hinder accurate weight measurement, or for which weight loss is contraindicated or could cause weight loss (e.g., cancer).
2. Current diagnosis of psychosis or bipolar disorder.
3. Unstable or recent onset of cardiovascular disease within 6 months or presence of congestive heart failure
4. Illness that might be associated with weight change, such as asthma (because of treatment with corticosteroids), psychosis
5. Use of medications that might cause weight gain such as hypoglycemic oral medicines or insulin, anti-depressants, and weight loss medications.
6. Unwilling or unable to provide informed consent.
7. Receiving disability insurance.
8. Pregnant or nursing in past 6 months, or plans to become pregnant within 12 months.
9. Enrolled in a weight loss program or study or member of household enrolled in study.
10. Residence outside of Marion County, Indiana.
11. Residence relocation plans within 12 months.
12. Planned or prior bariatric surgery.
13. Substance abuse.
14. History of treatment for eating disorder.
15. Unstable weight with loss or gain of ≥ 5% in last 3 months.

    -

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
BMI | two months

SECONDARY OUTCOMES:
2-Minute Step Test | two months
  Number of steps completed in two minutes
Chair stand test | 2 month

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O Clark, PhD., Principal Investigator — Indiana University Center for Aging
Locations (1):
- HITS, Indianapolis, Indiana, United States